CLINICAL TRIAL: NCT07203053
Title: A Multicentre Phase II Trial of Tarlatamab in Patients With Pretreated Extensive-stage Small Cell Lung Cancer (ES-SCLC) and ECOG PS 2
Brief Title: A Trial of Tarlatamab in Patients With Pretreated Extensive-stage Small Cell Lung Cancer (ES-SCLC) and ECOG PS 2
Acronym: START-lung
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 29-25
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Lung Small Cell Cancer
Keywords: ES-SCLC; Tarlatamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tarlatamab (Experimental)
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Protocol treatment consists of tarlatamab, administered as an intravenous (i.v.) infusion:
  * 1 mg on day 1 (C1D1),
  * 10 mg on day 8 (C1D8) and
  * 10 mg on day 15 (C1D15),
  * then 10 mg every two weeks (Q2W) until disease progression according to RECIST v1.1 criteria, unacceptable toxicity, or patient decision, whichever comes first.

SUMMARY:
START-lung is an international, multicentre, single-arm phase II trial. Protocol treatment consists of tarlatamab administered as an intravenous infusion until disease progression according to RECIST v1.1 criteria, unacceptable toxicity, or patient decision, whichever comes first. The primary objective of the trial is to assess the clinical efficacy of tarlatamab, in terms of 12-month OS rate, in patients with ES-SCLC and ECOG PS 2 who have previously received only one line of platinum-etoposide doublet chemotherapy with immune-checkpoint inhibition and whose disease has progressed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ES-SCLC.
* Previous treatment with only one line of platinum-etoposide doublet chemotherapy with immune-checkpoint inhibition for SCLC.

Patients treated with a platinum-etoposide doublet chemotherapy for prior limited stage (LS)-SCLC may be eligible for the study if the disease has progressed on treatment or within 6 months from chemotherapy completion (i.e. during durvalumab consolidation): the platinum-etoposide line of therapy will count as one prior line of therapy.

* Progressive disease on or after the first-line treatment for SCLC.
* ECOG Performance Status 2.
* Age ≥18 years.
* Adequate haematological, renal and liver function.
* Coagulation function: Prothrombin time (PT)/international normalised ratio (INR) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5x ULN, except for patients receiving anticoagulation, who must be on a stable dose of anticoagulation therapy for 6 weeks prior to enrolment.
* Pulmonary function:

  * No clinically significant pleural effusion. Pleural effusion managed with indwelling pleural catheter (e.g., PleurX) are allowed.
  * Baseline oxygen saturation >90% on room air.
* Cardiac function: Left ventricular ejection fraction (LVEF) ≥50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan (preferred), and no clinically significant electrocardiogram (ECG) findings.
* Women of childbearing potential, must have a negative urinary or serum pregnancy test within 5 weeks before enrolment. Pregnancy test must be repeated within 3 days before the first dose of tarlatamab treatment.
* Written Informed Consent must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

* Symptomatic CNS metastases Patients with untreated asymptomatic brain metastases and patients with treated and stable brain metastases are eligible.
* Diagnosis or evidence of leptomeningeal disease or spinal cord compression
* Prior history of immune-checkpoint inhibitor treatment resulting in:

  * any severe or life-threatening immune-mediated adverse event,
  * history of immune-mediated encephalitis or another immune-mediated CNS event (any grade),
  * grade ≥2 immune-mediated recurrent pneumonitis,
  * infusion-related reactions leading to permanent discontinuation of the immunotherapy agent.

Exception: patients with a history of immune-checkpoint inhibitor-induced endocrinopathy which is clinically stable on replacement therapy.

* Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
* History of solid organ transplantation.
* Treatment with live virus, including live-attenuated vaccination within 14 days prior to enrolment and inactive vaccines (e.g., non-live or non-replicating agent) and live viral non-replicating vaccines (e.g., Jynneos for Monkeypox infection) within 3 days prior to enrolment.
* History of other malignancy within the past 2 years, with the following exceptions:

  * Low-risk malignancy treated with curative intent and with no known active disease present for ≥1 year before enrolment and believed to be at low risk for recurrence per investigator discretion.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
  * Adequately treated breast ductal carcinoma in situ without evidence of disease.
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer.
  * Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association >class II) within 12 months prior to enrolment.
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 12 months prior to enrolment.
* Presence/history of an uncontrolled viral infection:

  * Known uncontrolled human immunodeficiency virus (HIV) infection.
  * Active hepatitis C infection (patients with detectable hepatitis C antibody [HCV Ab] and HCV RNA viral load above the limit of quantification).
  * Patients with presence of HCV Antibodies and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed.
  * Active hepatitis B infection (presence of hepatitis B surface antigen [HBsAg] and hepatitis B virus [HBV] DNA viral load above the limit of quantification [HBV DNA positive]).
  * Patients with resolved HBV infection defined as absence of HBsAg and presence of HBV core antibody (anti-HBc) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
  * Patients with chronic HBV infection inactive carrier state defined as presence of HBsAg and HBV DNA viral load below the limit of quantification [HBV DNA negative] are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
* Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to first dose of study treatment.

  * Prophylactic dexamethasone for the management of tarlatamab-related adverse events and any anti-emetic therapies are allowed.
  * Low-dose corticosteroids (prednisone ≤10 mg per day or equivalent) is permitted during the trial.
* Patients with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.

  * Patient has known active infection requiring parenteral antibiotic treatment. Upon completion of parenteral antibiotics and resolution of symptoms, the patient may be considered eligible for the study from an infection standpoint.
  * Note: Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment. Subjects requiring oral antibiotics who have been afebrile for >24 hours, have no leucocytosis, nor clinical signs of infection are eligible. Screening for chronic infectious conditions is not required unless otherwise noted as exclusion criteria.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Major surgical procedures within 5 weeks prior to enrolment.
* Any concurrent medical condition which, in the opinion of the investigator, would compromise patient safety or interfere with the evaluations for tarlatamab.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial until at least 60 days after the last dose of tarlatamab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate at 12 months (12-month OS) | OS is defined as the time from the date of enrolment until death from any cause. Assessed for approximately up to 41 months.
  The OS rate at 12 months is the primary endpoint of the trial. It is defined as the proportion of patients who are alive at 12 months from enrolment. The rate will be calculated as the number of patients alive at 12 months divided by the number of patients on follow-up at 12 months or with an earlier observed death event.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Assessed for approximately up to 41 months.
  Objective response rate (ORR) is defined as the rate of patients, among all those enrolled, who achieve a best overall response [complete response (CR) or partial response (PR)] according to the RECIST v1.1 across all post-enrolment time-points until the end of follow up for disease progression.
Duration of response (DoR) | Assessed for approximately up to 41 months.
  Duration of response (DoR) is defined as the time from the date of first documentation of objective response (CR or PR according to RECIST v1.1) to the date of first documented progression or death. Censoring will occur at the last tumour assessment with response other than progression. Patients without tumour assessment after documented objective response will be censored at the date of documented objective response (plus 1 day).
Disease control rate (DCR) | Assessed for approximately up to 41 months.
  Disease control rate (DCR) is defined as the rate of patients, among all those enrolled, who achieve CR or PR according to RECIST v1.1 or stabilisation of disease (SD), lasting for at least 12 weeks.
Progression-free survival (PFS) | Assessed for approximately up to 41 months.
  Progression-free survival (PFS) is defined as the time from the date of enrolment until documented progression (according to RECIST v1.1) or death if progression is not documented. Censoring (for patients without documented progression or death) will occur at the date of last tumour assessment. Patients without a post-baseline tumour assessment will be censored at the date of enrolment (plus 1 day).
Incidence, nature, and severity of adverse events | Assessed for approximately up to 41 months.
  Incidence, nature, and severity of adverse events according to CTCAE v5, except for CRS and ICANS, that are graded according to the ASTCT criteria21 and TLS that are graded according to the Cairo-Bishop classification
  All safety parameters will be summarised in tables to evaluate the toxicity/safety profile of the protocol treatment based on:
  * Adverse events (AEs) according to CTCAE v5.0 (any-cause as well as treatment-related) including AEs leading to dose delays and/or interruptions, withdrawal of protocol treatment, and death.
  * Occurrence of CRS and ICANS, defined according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria published by Lee et al. (2019).
  * Occurrence of TLS, defined according to the Cairo-Bishop classification.22
  * Severe and serious AEs.
  * Laboratory parameters and abnormalities, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Pérol, MD, Study Chair — Centre Léon Bérard, Lyon, France; Federico Capuzzo, MD, Study Chair — IRCCS Regina Elena, Rome, Italy
Locations (19):
- France (4):
  - CHU Angers, Angers
  - Institut Bergonie, Bordeaux
  - Lyon - Centre Léon Bérard, Lyon
  - Hôpital Nord de Marseille, Marseille
- Henry Dunant Hospital Center, Athens, Greece
- Italy (5):
  - Irccs Irst, Meldola
  - Instituto Europeo di Oncologia (IEO), Milan
  - Santa Maria della Misericordia Hospital, Perugia
  - AO San Giovanni Addolorata, Roma
  - Istituto Nazionale Tumori "Regina Elena", Roma
- Spain (5):
  - Hospital General Universitario Alicante, Alicante
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Hospital Universitatrio Vall d'Hebron, Barcelona
  - ICO Hospitalet H. Duran I Reynals / H. Bellvitge, Barcelona
  - Hospital Universitatrio Puerta del Hierro, Madrid
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - HFR - Hôpital cantonal, Fribourg
  - Geneva University Hospitals, Geneva
  - Kantonsspital St.Gallen, Sankt Gallen